CLINICAL TRIAL: NCT03253081
Title: Heterogeneity in ASD: Biological Mechanisms, Trajectories, and Treatment Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Connie Kasari, Ph.D., Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2P50HD055784-11 (NIH)
Record Dates: First submitted 2017-08-07; First posted 2017-08-17 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Children With Autism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PARENT focused intervention (Active Comparator): The PF condition will consist of a 90-minute parent group session twice per week. The group will comprise 3 to 4 parents and will focus on psychoeducation and support/well-being for the parent.
  Interventions: Behavioral: PARENT focused intervention
- CHILD focused intervention (Active Comparator): In the CF condition both parent and child will attend the 90-minute session twice weekly. The session will be divided into 30-minute segments and include two 30-minute individualized 1-on-1 sessions with a trained interventionist.
  Interventions: Behavioral: CHILD focused intervention

INTERVENTIONS:
Behavioral: PARENT focused intervention — The group will comprise 3 to 4 parents and will focus on psychoeducation and support/well-being for the parent. Sessions will include a 20-minute welcome and supportive discussion where parents can provide updates on their week and seek advice and support from the group, followed by a 45-minute interactive education session focused on the principles of JASPER, and close with a 20-minute Mindfulness session. The Mindfulness session will be led by a certified expert.
  Arms: PARENT focused intervention
Behavioral: CHILD focused intervention — The session will be divided into 30-minute segments and include two 30-minute individualized 1-on-1 sessions with a trained interventionist. One of these two sessions will involve the parent in hands-on training while the other will be interventionist-led while the parent observes. The remaining 30-minutes will include a snack for the child and time for the parent to discuss and ask questions of the interventionist regarding the session content.
  Arms: CHILD focused intervention

SUMMARY:
Parent-mediated interventions often target social communication in young children with ASD, although to date studies yield inconsistent effects. One reason for the limited evidence may be the considerable heterogeneity in both parent and child characteristics that affect the fit of intervention to family and ultimately influence treatment outcome. For parents, these factors might include stress associated with the uncertainty of their child's diagnosis, caregiver expectations for the intervention itself, and a parent's own style of interaction that may be influenced by milder but qualitatively similar ASD characteristics, known as the broad autism phenotype (BAP). For children, these factors might include nonverbal DQ, language, or sensory impairment. The fit between type of intervention and optimal outcome for parent and child is an understudied, yet essential component of early intervention that may be susceptible to the influence of heterogeneity in the parent and child. One approach to addressing this variability is to implement an adaptive intervention approach that seeks to capitalize on heterogeneity among children and parents. Utilizing an adaptive treatment design, the current study tests the optimal sequence of intervention delivery and specific parent and child characteristics that may moderate treatment success in three 10-week stages of intervention. The first phase will randomize parents and children to a parent education condition, consisting of a parent support and education group focused on social communication development, or to a parent mediated and therapist delivered condition involving coaching of the parent with their child in social communication strategies. Phase 2 involves re-randomizing parents and children to maintain the same treatment arm, or change to the opposite arm to test the optimal sequence of intervention delivery and specific parent and child characteristics that may moderate treatment success. In the final phase, dyads are randomized to different maintenance arms, each comprised of 5 sessions with one involving skype and text contact, the other in -home visits, to explore how best to maintain treatment gains once the active intervention phase is complete. This study has the potential to dramatically improve child social communication outcomes by individualizing and personalizing parent intervention approaches with very young children, a high priority need of the Interagency Autism Coordinating Council and NIH.

DETAILED DESCRIPTION:
While social communication is a core developmental deficit that characterizes children with ASD, there is great heterogeneity in both presentation and gains with treatment. Long term outcomes of children with ASD vary with nearly 40% remaining minimally verbal by school age. Beginning early and providing high doses of intervention appears critical to child outcomes, and one cost-effective, efficient way to accomplish these goals is to involve parents. Particularly, for very young children (under the age of 3 years) who may not have a confirmed ASD diagnosis, parent mediated interventions have several advantages. One is that there is potential for earlier access to evidence based interventions. Parents can intervene with their child immediately without waiting for access through a lengthy diagnostic process or for therapist -delivered interventions that can have long wait times. Another is that parents can increase the dose of an intervention since they are with their child for many more hours than non-family members.

Despite the increasing numbers of parent mediated interventions, inconsistent results are noted. A few studies have found significant differences in both child and parent outcomes but others find limited to no effects on parent and/or child. This heterogeneity in outcomes is often attributed to child characteristics or to the intervention itself. However, the fit between type of intervention-focused on the parent-(education about social communication in their child, or stress reduction interventions), or focused on the child-(parent coached to work directly with their child)-has rarely been examined in parents engaged in these interventions. Fit may be influenced by parent characteristics that can affect their ability to implement the interventions.

These include stress associated with the uncertainty of their child's diagnosis, caregiver expectations for the intervention itself, and parent's own style of interaction that may be influenced by milder but qualitatively similar ASD characteristics, known as the broad autism phenotype.

It is widely recognized that a single intervention is not effective for all parents and children. One approach to addressing this variability is to implement an adaptive intervention approach that seeks to capitalize on heterogeneity and evolving status among children and parents. An adaptive intervention is a replicable, sequence of treatment decision rules designed to help guide clinicians concerning whether, how or when-and based on which measures-to provide certain intervention components. This type of intervention design provides information on the most effective intervention for children and parents who need it (leading to individualized and personalized sequences of treatment). Using a novel experimental design, the proposed study will develop a more effective adaptive intervention by addressing the following specific aims:

Primary Aim (Best Initial Strategy): To determine the effect of PARENT focused intervention vs CHILD focused intervention on change in child initiated joint engagement (primary outcome), play, and joint attention (secondary outcomes) from baseline to end of phase 1. Hypothesis: Children will improve more, on average, when offered CHILD focused intervention.

Secondary Aim 1 (Best Sequence): To compare and contrast the four pre-specified adaptive interventions from baseline to end of phase 2 on primary and secondary outcomes. Hypothesis: The sequential intervention beginning with CHILD focused interventions followed by PARENT education sessions will lead to the most improved outcomes.

Secondary Aim 2 (Toward More Personalized Intervention Sequences): To develop a more individually- tailored adaptive intervention by examining whether parental factors including BAP, parental stress, or parent's expectancies for the intervention, and child factors including non-verbal DQ, language or sensory impairment at baseline moderates the effect of Phase 1 interventions from baseline to end of Phase 1 on primary and secondary outcomes. Hypotheses: (i) Children with parents who report greater BAP and parenting stress will benefit more from PARENT focused intervention and children with parents who report greater expectancy will benefit more from CHILD focused intervention. (ii) Children with low non-verbal DQ and high levels of sensory impairment at baseline will benefit more from the CHILD focused intervention from baseline to end of phase 1. Secondary Aim 3 (Maintenance Protocol): To determine the maintenance effect of in person home visits versus technology supported maintenance protocol on change in primary and secondary outcomes from (i) baseline to end of phase 3 and (ii) from end of phase 2 to end of phase 3. Hypothesis: Children in the home visit maintenance protocol will have more improved outcomes from baseline to end of phase 3 compared to the children in the technology supported maintenance protocol.

Secondary Aim 4 (Exploratory: Biomarkers and Genetics): To characterize children at risk of ASD in terms of electrophysiological biomarkers (neural synchrony measured by EEG power, peak alpha frequency and coherence) and genetic risk (as measured by the presence of CNVs and polygenetic risk score) and to explore each's role as a biological moderator of treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Have elevated scores on the ADOS-2 and clinical concern from a professional (Pediatrician, Psychologist, etc.). For children under the age of 30 months, some of whom may not have a diagnosis of ASD, they must show elevated risk in the mild-to-moderate or moderate-to-severe risk categories on the ADOS-T. For children over the age of 30 months, they must meet clinical cutoff on the ADOS-2, Module 1 or 2.

  * Are between 12 months and 36 months
  * Have a parent available for parent-mediated sessions 2 times per week in the classroom

Exclusion Criteria:

* Do not have seizures or are stable on anti-seizure medication

  * Do not have associated physical disorders
  * Are not co-morbid with other syndromes or diseases unless they come from Project I in our center- 22q11 deletion or TSC children at 12 months with concern for ASD on the ADOS-T.

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Joint Engagement on the Caregiver-child interaction (CCX) over the course of the study | Baseline(entry), Phase1 midpoint (5 weeks post entry) and end(10 weeks post entry), Phase2 midpoint (15 weeks post entry) and end(20 weeks post entry), and Phase3 midpoint(25 weeks post entry) and end(30 weeks post entry), and 1 year follow-up post entry
  A 10-minute interaction between parent and child. These sessions will be carried out with a standard set of toys and videotaped.
  Parents will be asked to engage their child in play as usual. Coders blind to child treatment assignment and time point will code the videotapes according to Adamson et al, 2004 coding procedures, the same as used in our previous studies (Harris, Kasari, & Sigman, 1996; Kasari et al, 2006; Kasari, et al, 2008). Joint engagement change will be recorded and measured throughout the study.

SECONDARY OUTCOMES:
Early Social- Communication Scales | Baseline(entry), Phase 1 end(10 weeks post entry), Phase 2 end(20 weeks post entry), Phase 3 end(30 weeks post entry), and 1 year follow-up post entry
  In this semi-structured interaction, the child and tester sit facing each other at a table with a set of toys in view but out of reach of the child which are introduced one by one (Mundy, Sigman, Ungerer, & Sherman, 1986; Seibert, Hogan, & Mundy, 1982).
The Structured Play Assessment-R | Baseline(entry), Phase 1 end(10 weeks post entry), Phase 2 end (20 weeks post entry), Phase 3 end (30 weeks post entry), and 1 year follow-up post entry
  SPA-R is designed to obtain the child's highest levels of spontaneous play acts. The child is presented with 5 different play sets by the experimenter; the entire play interaction last about 15-20 minutes. The child's play behaviors are videotaped and later coded. The variables of interest include the frequency of child initiated functional and symbolic play acts and also the count of different novel types of acts. This measure has shown excellent reliability and validity across a range of studies (Kasari et al., 2006; Sigman & Ruskin, 1999; Sigman & Ungerer, 1984).
Parenting Stress Index (PSI) | Baseline(entry), Phase 1 end(10 weeks post entry), Phase 2 end(20 weeks post entry), Phase 3 end(30 weeks post entry), and 1 year follow-up post entry
  total parental stress
The Broader Autism Phenotype Questionnaire (BAPQ) | Baseline (entry)
  score comprised of three subscales: aloof, rigid and pragmatic language.
Caregiver Expectancies /Belief in the Intervention | Baseline (entry)
  This measure (Nock & Kazdin, 2001) assesses parent's beliefs about whether the intervention is appropriate and working for his/her child. It reflects the parent's motivation to participate, their belief in the intervention's value, and its effectiveness. Scoring of the measure consists of a series of ratings on a Likert scale summed to obtain a total score.
BOSCC | Baseline(entry), Phase 1 mid(5 weeks post entry) and end(10 weeks post entry); Phase 2 mid (15 weeks post entry) and end(20 weeks post entry); Phase 3 mid (25 weeks post entry) and end (30 weeks post entry) and I year follow up post entry
  Social Communication Total Score
Caregiver-child interaction (CCX) | Baseline (entry), Phase 1 end (10 weeks post entry), Phase 2 end (20 weeks post entry), Phase 3 end (30 weeks post entry), and 1 year follow-up post entry
  A 10-minute interaction between parent and child. These sessions will be carried out with a standard set of toys and videotaped.
  Parents will be asked to engage their child in play as usual. Coders blind to child treatment assignment and time point will code the videotapes according to Adamson et al, 2004 coding procedures, the same as used in our previous studies (Harris, Kasari, & Sigman, 1996; Kasari et al, 2006; Kasari, et al, 2008). Change will be recorded and measured throughout the study for joint attention and play.

OTHER OUTCOMES:
Nonverbal Developmental Quotients (DQ) from Mullen | Baseline
  Nonverbal Development Quotients (DQ) (DQ; mental age ÷ chronological age)
An electroencephalogram (EEG) test | Baseline
  EEG
Presence of copy-number variations (CNVs) | Baseline
  DNA
Polygenetic risk score (PRS) | Baseline
  DNA
Sensory Impairment from ITSP | Baseline
  Sensory impairment score

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States